Official title: Which Physical Therapy Program is Cost-effective in Knee Osteoarthritis?

NCT number: NCT04736069 document date: 3.10.2010

**Informed Consent Form** 

**Title of the Study:** Which Physical Therapy Program is Cost-effective in Knee Osteoarthritis?

**Volunteer Number:** 

**Initials of the Volunteer's Name:** 

"You are invited to a scientific study. Before making your decision, it is important to understand what will be done in this research and why. Please read the explanations below carefully. If you wish, discuss it with your friends, family and doctor. Ask us if there are any unclear points or if you want further clarification. Think carefully about whether to participate in this research."

Knee osteoarthritis (OA) increases with age. Education, medical treatment methods, physical therapy applications, exercise, orthosis-prosthesis, shoe modifications (such as lateral wedge, knee brace) are used in the treatment of knee OA. These applications can be applied on an outpatient or hospital basis. This diversity also changes treatment costs. In this study, it was aimed to compare the effectiveness of outpatient and inpatient physical therapy applications, exercise and lateral wedge applications on shoes on pain, mobility, functionality and quality of life, and the long-term cost-effectiveness of these applications in patients with knee osteoarthritis. The reason we include you in this study is that you also have knee osteoarthritis.

If you participate in this study, your knee will be evaluated by physical examination. Your pain will be evaluated with the pain rating scale and you will be questioned with 3 different questionnaires to investigate the effects of your pain on your quality of life and functional capacity. Your range of motion will be measured during physical examination. Some tests will be done to measure your functional capacity (100 meters walking time, time to climb stairs, time to sit and get up from a chair). These measurements won't hurt you. Your diagnostic blood tests, knee film, and magnetic resonance imaging or computed tomography will be performed. These are necessary for your diagnosis. The fees for these will be collected from your health institution. These examinations are the routine tests we order for your diagnosis and to consider treatment options; not that because you have been included in this study. Physical therapy applications performed during your treatment and follow-up, if necessary, injection, medication, medical equipment such as knee brace, loss of work day due to knee pain in post-treatment follow-up, need to see a doctor again, have an examination or physical therapy, balneotherapy or alternative treatment needs, and costs will be asked. Your evaluation will be done 5 times before, after treatment, in the 1st, 3rd and 6th months. No difference fee will be charged from the applied physical therapy, and the treatment fee paid by your health institution will be charged. No difference will be requested from the inspection.

60 patients with knee osteoarthritis like you will participate in the study and will be divided into 2 groups. Which group you will be in will be determined according to the card you take from the closed envelope. One of the groups will be applied for 3 weeks, 5 days a week, 45 minutes of physical therapy equipment (superficial hot packs and ultrasound as deep warming) and pain relief current (TENS) inpatient and exercise program will be given to strengthen the muscles around the knee. In the second group, for 3 weeks, 5 days a week, 45 minutes of physical therapy equipment, hot treatment (superficial hot packs and ultrasound as deep warming) and pain relief current (TENS) will be applied and a home exercise program will be given. Our aim is to compare the midlong term cost effectiveness of these applications.

You do not have to participate in this study. If you do not want to participate in this study, the necessary treatments for your illness will be still applied. You will not be paid for participating in the study. You will not be asked to pay extra money. You will not be excluded from the study against your will. If only you do not attend the treatment regularly and if you skip days, you will be excluded from the study by the researcher. If you want to agree to participate in the study and leave later, you can quit. Your necessary treatments will continue as they are. All your personal information in this study will be kept confidential. Only your doctor will know. If there is any development during the investigation that may be of interest to you, you will be notified immediately or immediately to your legal representative. This study will be done with the approval of the ethics committee."If I want to get more information or there is an emergency, I can call my doctor.""It is possible to consult your doctor for more information about the study and in case of any side effects that may occur during the treatment.

For information, You can contact Prof. Dr. Deniz Evcik directly or call 2044262. "

I have read the information form regarding the above study. I was able to ask the questions I had in mind. I understood that my participation in this research was on a voluntary basis. If I want, I can decide to withdraw from this study without giving any reason and without disrupting my subsequent medical care. I understand that my medical records will be reviewed by the health authorities, and I allow these people. Under these conditions, I agree to participate in the study of my own free will without any pressure or coercion.

A copy of this form has been given to me for re-reading and obtaining information if required.

## Participant Name and surname:

Address:

Phone Signature

## **Interview witness Name and surname:**

Address: Phone. Signature:

## The physician meeting with the participant Name, surname, title:

Phone.

Signature: Address: